CLINICAL TRIAL: NCT04904679
Title: The Use of Amniotic Membrane or Inverted Internal Limiting Membrane Flap for Large or Refractory Macular Holes: a Prospective, Comparative Study Using Microperimetry
Brief Title: The Use of Amniotic Membrane or Internal Limiting Membrane for Large or Refractory Macular Holes: A Prospective Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Oftalmologico de Sorocaba (Other)
Responsible Party: Principal Investigator, Anna Carolina Carvalho Araujo, Ophthalmologist , MD, Hospital Oftalmologico de Sorocaba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAMprotocol
Record Dates: First submitted 2021-05-17; First posted 2021-05-27 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Macular Holes
Keywords: Human Amniotic Membranes in macular holes using microperimetry
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, unmasked single center interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniotic Membrane group (Active Comparator): Patients who will be treated with a amniotic membrane plug
  Interventions: Device: Pars plana Vitrectomy with internal limiting membrane peeling
- Internal Limiting Membrane group (Active Comparator): patients who will be treated with a internal limiting membrane flap
  Interventions: Device: Pars plana Vitrectomy with internal limiting membrane peeling

INTERVENTIONS:
Device: Pars plana Vitrectomy with internal limiting membrane peeling — The pars plana 23-gauge (23G) vitrectomy technique will be performed with removal of the internal limiting membrane (ILM) (when adhered to the macula) and placement of either an amniotic membrane plug or an ILM flap in the macular hole. This will be followed by a fluid-air exchange and buffering gas infusion (12.5% C3F8).
  The amniotic membrane plug will be prepared using a dermatological punch with a diameter of 1 to 2 mm, depending on the size of the macular hole as measured by OCT. It will be positioned inside the macular hole using 23G forceps, with its chorionic side facing the retinal pigmented epithelium (RPE).
  The ILM flap will be created at the time of peeling-with an inverted flap in primary cases and a free flap in refractory cases. It will be positioned over the hole (inverted flap) or inside the macular hole (free flap) using 23G ILM forceps.
  These techniques will be assisted by the use of an extra lighting sclerotomy.
  Other Names: Use of Amniotic membrane plug; Use of a internal limiting membrane inverted flap; gas tamponade (C3F8 12,5%)

SUMMARY:
Prospective, randomized, unmasked interventional study. To evaluate anatomical and functional results through microperimetry in cases of refractory or large macular holes (MH), using amniotic membrane (AM) or internal limiting membrane ( ILM ).

DETAILED DESCRIPTION:
This study will evaluate functional outcomes through microperimetry in patients undergoing macular hole surgery. It will focus on patients with macular holes ≥600 microns, as well as those with holes refractory to conventional surgical treatment. The study will assess the use of amniotic membrane or internal limiting membrane (ILM) as adjuncts in the macular hole closure process.

The gold-standard treatment for idiopathic macular holes is pars plana vitrectomy (PPV), which involves removal of the posterior hyaloid (when adhered) and the ILM using a vital dye, followed by placement of buffering gas (C3F8 or SF6) at a non-expandable concentration. However, approximately 44% of large macular holes remain unclosed after conventional surgery.

To improve closure rates in such cases, new techniques have been introduced, including the inverted ILM flap technique and the free ILM flap technique. While studies demonstrate the effectiveness of these techniques, they show no significant improvement in visual function.

The amniotic membrane (AM) has recently been explored as an adjunct for macular hole closure and as a substrate for cell growth and visual acuity improvement. Amniotic membranes are believed to promote epithelialization and possess anti-fibrotic, anti-inflammatory, anti-angiogenic, and antimicrobial properties.

In this study, eligible patients will be randomized into two groups:

* Group 1: Undergoing PPV with ILM removal, followed by placement of an amniotic membrane plug inside the macular hole, with its chorionic face in contact with the retinal pigment epithelium (RPE).
* Group 2: Undergoing PPV with ILM removal, followed by placement of either an inverted ILM flap or a free ILM fragment for refractory cases, positioned over (inverted flap) or inside (free flap) the macular hole.

Once the AM plug or ILM flap is confirmed in its correct location, a fluid-gas exchange will be performed with 12.5% C3F8 buffering gas, and patients will maintain a face-down position for 7 days postoperatively.

Patients included in the study will undergo:

* Preoperative assessment, including best-corrected visual acuity (BCVA) measurement, optical coherence tomography (OCT) using the Zeiss Cirrus 5000, and microperimetry using the Macular Integrity Assessment (MAIA) device.
* Postoperative evaluations at day 1 and day 7, followed by assessments at 1, 3, 6, and 12 months. During these visits:- A complete ophthalmic examination will be performed.
* OCT imaging will be conducted at day 7, month 1, month 3, month 6, and month 12.
* Microperimetry will be conducted at months 1, 3, 6, and 12 to evaluate anatomical and functional responses.

The use of the amniotic membrane, given its anti-inflammatory, anti-fibrotic, and cell growth-supporting properties, is expected to increase closure rates in refractory and large macular holes and contribute to better functional outcomes by supporting outer retinal layer regeneration.

The Sorocaba Eye Bank (BOS) will provide, prepare, and preserve the amniotic membrane used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a macula hole that falls into the two categories below:
* Patients with idiopathic macular hole (with no history of secondary macular hole) ≥ 600 microns (measured using optical coherence tomography)
* Patients with an idiopathic macular hole submitted to conventional treatment without closing it (of any size).
* History of the disease less than 18 months
* Aged over 18 years old
* Visual acuity less than 20/32

Exclusion Criteria:

* History of any previous macular disease other than idiopathic macular hole
* Macular hole of other causes (secondary)
* Patients with diabetic retinopathy or other retinal vascular diseases
* Eyes subjected to intravitreal injection of any medication
* Visual acuity <20/400 of any retinal cause in the contralateral eye or absence of the globe *Aged under 50 years old
* Cataract and anti-glaucoma surgery less than 3 months before the study
* Glaucoma with optic nerve excavation > 0.7 in the studied eye
* Intraocular pressure > 24 mmHg with the use of maximum medication in the studied eye
* History of vitreoretinal surgery for a condition other than the idiopathic macular hole (retinal detachment, vitreous hemorrhage)
* History of retinal detachment of any etiology
* A patient who manifests himself not being able to perform the head position in the postoperative period
* A patient with active anterior or posterior uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The retinal sensitivity | through study completion, an average of 1 year
  measured by the microperimetry
The fixation stability | through study completion, an average of 1 year
  measured by the microperimetry

SECONDARY OUTCOMES:
the macula hole closure rate | through study completion, an average of 1 year
  measured by OCT

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital Oftalmologico de Sorocaba/ Banco de Olhos de Sorocaba, Sorocaba, São Paulo
  - Sorocaba Eye's Hospital, Sorocaba, São Paulo

IPD SHARING:
Plan to Share IPD: No
Only the microperimetry graphs and OCT images will be published, without any IPD.

REFERENCES:
- [Result] Jirsova K, Jones GLA. Amniotic membrane in ophthalmology: properties, preparation, storage and indications for grafting-a review. Cell Tissue Bank. 2017 Jun;18(2):193-204. doi: 10.1007/s10561-017-9618-5. Epub 2017 Mar 2. PMID 28255771
- [Result] Ferreira MA, Maia A, Machado AJ, Ferreira REA, Hagemann LF, Junior PHER, Rezende FA. Human amniotic membrane for the treatment of large and refractory macular holes: a retrospective, multicentric, interventional study. Int J Retina Vitreous. 2021 May 8;7(1):38. doi: 10.1186/s40942-021-00308-6. PMID 33964971
- [Result] Caporossi T, Tartaro R, De Angelis L, Pacini B, Rizzo S. A human amniotic membrane plug to repair retinal detachment associated with large macular tear. Acta Ophthalmol. 2019 Dec;97(8):821-823. doi: 10.1111/aos.14109. Epub 2019 Apr 6. PMID 30953398
- [Result] Rizzo S, Caporossi T, Tartaro R, Finocchio L, Franco F, Barca F, Giansanti F. A Human Amniotic Membrane Plug to Promote Retinal Breaks Repair and Recurrent Macular Hole Closure. Retina. 2019 Oct;39 Suppl 1:S95-S103. doi: 10.1097/IAE.0000000000002320. No abstract available. PMID 30312261
- [Result] Caporossi T, Pacini B, De Angelis L, Barca F, Peiretti E, Rizzo S. HUMAN AMNIOTIC MEMBRANE TO CLOSE RECURRENT, HIGH MYOPIC MACULAR HOLES IN PATHOLOGIC MYOPIA WITH AXIAL LENGTH OF >/=30 mm. Retina. 2020 Oct;40(10):1946-1954. doi: 10.1097/IAE.0000000000002699. PMID 31868775
- [Result] Meyer CH, Borny R, Horchi N. Subretinal fluid application to close a refractory full thickness macular hole. Int J Retina Vitreous. 2017 Nov 27;3:44. doi: 10.1186/s40942-017-0094-7. eCollection 2017. PMID 29209516
- [Result] Kase S, Saito W, Mori S, Saito M, Ando R, Dong Z, Suzuki T, Noda K, Ishida S. Clinical and histological evaluation of large macular hole surgery using the inverted internal limiting membrane flap technique. Clin Ophthalmol. 2016 Dec 16;11:9-14. doi: 10.2147/OPTH.S119762. eCollection 2017. PMID 28031697
- [Result] Ch'ng SW, Patton N, Ahmed M, Ivanova T, Baumann C, Charles S, Jalil A. The Manchester Large Macular Hole Study: Is it Time to Reclassify Large Macular Holes? Am J Ophthalmol. 2018 Nov;195:36-42. doi: 10.1016/j.ajo.2018.07.027. Epub 2018 Jul 30. PMID 30071212
- [Result] Passemard M, Yakoubi Y, Muselier A, Hubert I, Guillaubey A, Bron AM, Berrod JP, Creuzot-Garcher C. Long-term outcome of idiopathic macular hole surgery. Am J Ophthalmol. 2010 Jan;149(1):120-6. doi: 10.1016/j.ajo.2009.08.003. Epub 2009 Oct 20. PMID 19846059
- [Result] Lois N, Burr J, Norrie J, Vale L, Cook J, McDonald A, Boachie C, Ternent L, McPherson G; Full-thickness Macular Hole and Internal Limiting Membrane Peeling Study (FILMS) Group. Internal limiting membrane peeling versus no peeling for idiopathic full-thickness macular hole: a pragmatic randomized controlled trial. Invest Ophthalmol Vis Sci. 2011 Mar 1;52(3):1586-92. doi: 10.1167/iovs.10-6287. PMID 21051731
- [Derived] Carvalho Araujo AC, Bordon AF, Falcao V, Bortolai P, Dib E, Maia M. The use of amniotic membrane or inverted internal limiting membrane flap for large or refractory macular holes: a prospective, comparative study using microperimetry. Graefes Arch Clin Exp Ophthalmol. 2025 Sep 15. doi: 10.1007/s00417-025-06917-3. Online ahead of print. PMID 40952489